CLINICAL TRIAL: NCT02041559
Title: The Effect of Different Doses of Remifentanil on Kidney Function During Robot Assisted Prostatectomy - A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0753
Record Dates: First submitted 2014-01-13; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- robot assisted prostatectomy: robot assisted prostatectomy

SUMMARY:
Robot assisted prostatectomy reduces the patients' postoperative pain and leads to rapid rehabilitation. But pneumoperitoneum affects the kidney. The increase of stress hormone reduces the glomerular filtration and the vaso-contraction of renal vessels leads the renal ischemia. Remifentanil is analgesics coupled with μ opioid receptor. In high dose of remifentanil, it is associated with κ and δ receptors, which leads to renal protection effect in animal study. Also, remifentanil infusion during anesthesia showed a diuretic effect. The purpose of this study is to investigate the remifentanil effect on renal function during robot assisted prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* ages > 19 years and < 85 years
* the patients undergoing a general anesthesia for robot assisted prostatectomy

Exclusion Criteria:

* incomplete record
* history of opioid or steroid using
* solitary kidney
* history of kidney transplantation

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male patients undergoing robot assisted prostatectomy
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury incidence based on Acute Kidney Injury Network criteria | 24 hours after end of surgery
  Acute kidney injury incidence based on Acute Kidney Injury Network criteria was defined as increase in serum creatinine from baseline of ≥ 0.3 mg/dl within a 48-hour period. Acute kidney injury is evaluated at POD 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System, Seoul, South Korea